CLINICAL TRIAL: NCT02892357
Title: Efficacy of Traditional Chinese Medicine Jianpi Qinghua Granule Combined With Low Dose Omeprazole in Patients With Non-erosive Reflux Disease (NERD)
Brief Title: Efficacy of Traditional Chinese Medicine Combined With Omeprazole in Patients With Non-erosive Reflux Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Digestion-04
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2019-08-26 (Actual); Status verified 2019-02

CONDITIONS: Non-erosive Reflux Disease
MeSH Terms: conditions — Non-Erosive Reflux Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Participants in this group take the herbal compound of Jianpi Qinghua granules and half-dose omeprazole tablet.Jianpi Qinghua granule:one bag after 1 hour of breakfast and supper(twice a day) for 4 weeks.Half-dose omeprazole tablet:1 tablet of real omeprazole (10mg) and 1 tablet of Sham(10mg),once a day before breakfast for 4 weeks.
  Interventions: Drug: Treatment group
- Control group (Active Comparator): Participants in this group take the sham herbal granules twice a day as treatment group and two pieces of real omeprazole tablet(10mg each) once a day before breakfast for 4 weeks.
  Interventions: Drug: Control group

INTERVENTIONS:
Drug: Treatment group — Jianpi Qinghua granules:twice a day,1 bag a time;10mg omeprazole and 10mg sham ,once a day,all for 4 weeks.
  Other Names: Experimental group
  Arms: Treatment group
Drug: Control group — sham Jianpi Qinghua granules:twice a day,1 bag a time; 20mg omeprazole once a day ,all for 4 weeks.
  Other Names: Omeprazole group
  Arms: Control group

SUMMARY:
This is a double-blind,randomised,placebo-controlled clinical trial.We would like to investigate the safety and efficacy of Jianpi Qinghua granule(a Chinese herbal compound) combined with half-dose omeprazole in treatment of non-erosive reflux disease(NERD).

DETAILED DESCRIPTION:
This is a double-blind,randomised,placebo-controlled clinical trial.We recruit patients that suffer from non-erosive reflux disease and then divide them into two groups:treatment group and control group.Treatment group take Jianpi Qinghua granule and half-dose omeprazole for 4 weeks,control group take a normal dose of omeprazole for 4 weeks.Finally we investigate the safety of Jianpi Qinghua granule combined with half-dose omeprazole in treatment of non-erosive reflux disease(NERD),and contrast the efficacy of Jianpi Qinghua granule with omeprazole.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 18 and 75 years, able to read and write Chinese;
* Meet the criteria of diagnosis of NERD
* GERD Q score>=8
* Meet the TCM diagnosis of syndrome of dampness-heat due to spleen deficiency
* Receiving no other treatments during the study;
* Voluntarily agreeing with the study protocol and signing a written informed consent.

Exclusion Criteria:

* Gastro-duodenal ulcer
* Infections, inflammations, or obstruction of the small or large intestine
* History of gastrointestinal cancer, or prior surgery of the stomach or intestine
* Females who are pregnant or those lacking adequate contraception
* Unwilling to sign the informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-09 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of GERD Q Scale | 6 weeks
  GerdQ was developed through the integration of validated questionnaires reflecting psychological problems and the data of diagnoses of GERD in primary and secondary medical institutions. GerdQ is used for the diagnosis and management of GERD with good authenticity and reliability. GerdQ has six items: heartburn, regurgitation, abdominal pain, nausea, sleep disorders and use of OTC medications. The score is evaluated according to the frequency of every item occurred in recent one week. 0 day, 1 day, 2-3 days, 4-7days respectively assessed to the score of 0, 1, 2 and 3 in the items of heartburn, regurgitation, sleep disorders and use of OTC medications. 0 day, 1 day, 2-3 days, 4-7days respectively assessed to the score of 3, 2, 1 and 0 in the items of abdominal pain and nausea.

SECONDARY OUTCOMES:
Change of TCM Syndrome Questionnaire | 6 weeks
  The scale is based on the Clinical Guideline of New Drugs for Traditional Chinese Medicine. It is uesd to evaluate the discomfort of gastrointestinal system based on TCM theory. It contains 15 items of TCM terminology which used to assess severity of physical discomfort (0 = absent; 1 = mild; 2 = moderate; 3 = severe). The main concerns of these items include stomach distension, stomachache, appetite decrease, heartburn, acid regurgitation, sputum increase, feeling of obstruction in pharynx, feeling thirsty but not want water, feeling of distention on both sides of the lower abdomen, limbs weakness, short of breath, feeling weak and unwilling to speak, somatosensory heaviness, feeling afraid of the cold and having loose stool.
Change of 36-Item Short Form Survey Instrument(SF-36) | 6 weeks
  SF-36 reflects healthy condition.
Change of Patients Report Clinical Outcomes(PRO) | 6 weeks
  The PRO was developed by the digestive department of Xiyuan hospital. Considering the clinical characteristics of patients with chronic gastrointestinal diseases in China, we have spended two years to collect measurement indicators, screen and optimizing items, implement pre-survey of small samples and field survey, and finally formulated this current PRO. It contains 35 items in six dimensions (regurgitation, dyspepsia, physical status, ability to life, defecation situation and mental state). Our analysis of 274 questionnaires show that the PRO has good reliability and validity in reflecting the situation of chronic gastrointestinal diseases. Every item in PRO has five levels of discomfort(never, occasionally, sometimes, often, always) and they respectively represent the score of 0, 1, 2, 3 and 4.
Change of the Hamilton Depression Scale 17 item (HAMD17) | 6 weeks
  The scoring criteria of the scale were :(0)none;(1)mild;(2)moderate;(3)severe;(4) extremely heavy.A few items use the 3-grade scoring method with 0-2 points, and the grading standard is :(0) none;(1) mild to moderate;(2) severely.
Safety outcomes | 6 weeks
  Safty indexs contain adverse event, general medical examination, blood biochemical examination, urine and stool routine test and electrocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: fengyun Wang, Ph.D, Study Chair — xi yuan hospital
Locations (2):
- China (2):
  - Dongfang Hospital, Beijing, Beijing Municipality
  - Guanganmen Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Che H, Zhang B, Zhang C, Zhou B, Ji H, Xie J, Shi X, Li X, Wang F, Tang X. JianpiQinghua granule reduced PPI dosage in patients with nonerosive reflux disease: A multicenter, randomized, double-blind, double-dummy, noninferiority study. Phytomedicine. 2021 Jul 15;88:153584. doi: 10.1016/j.phymed.2021.153584. Epub 2021 May 3. PMID 34119741